CLINICAL TRIAL: NCT06487585
Title: Angiotensin II as First-Line Vasopressor Therapy in Cardiac Surgery (ANG-First Trial)
Brief Title: ANG-First Trial (Angiotensin II as First-Line Vasopressor Therapy in Cardiac Surgery)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland St. Joseph Medical Center (Other)
Collaborators: La Jolla Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00109542
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Vasodilatory Hypotension During or After Cardiac Surgery
Keywords: Vasodilation; Hypotension; Cardiopulmonary Bypass; Cardiac Surgery
MeSH Terms: conditions — Aneurysm; Hypotension | interventions — Angiotensin II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study Drug Arm - Angiotensin II arm (Other): Angiotensin II
  Interventions: Drug: Angiotensin II

INTERVENTIONS:
Drug: Angiotensin II — Angiotensin II: Starting dose of 2.5 ng/kg/min administered IV; may dose escalate up to 80 ng/kg/min in order to achieve a MAP of 65 mmHg or higher in the first 3 hours. After 3 hours, may escalate dose up to 40 ng/kg/min in order to achieve a MAP of 65 mmHg. Dose titration in increments of 10 ng/kg/min every 2 minutes.

SUMMARY:
The purpose of this research is to evaluate the use of Angiotensin II in patients with low blood pressure post-surgery. Your information will be collected for 28 days post the procedure and initiation of the study drug to assess for safety events and complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age undergoing cardiac surgery requiring CPB
* Patients must have clinical features of vasodilation as determined by a MAP < 65 mmHg that is non-transient in the opinion of the treating physician
* Patients must be adequately volume resuscitated in the opinion of the treating physician
* Systemic Vascular Resistance index (SVRi) < 1970 dynes·sec/cm⁵/m² to support the clinical diagnosis of vasodilation; if no pulmonary artery catheter is in place, vasodilatory hypotension diagnosis according to the judgement of the critical care team
* Biventricular systolic function is at or greater than pre-cardiopulmonary bypass baseline as demonstrated by echocardiographic evaluation, or the patient is concomitantly treated with

Exclusion Criteria:

* Bleeding as primary etiology of hypotension, as determined by > 4 units RBC transfusion in 24 hours.
* Patients on ECMO
* Patients with active endocarditis
* Patients already on renal replacement therapy or creatinine of > 4 mg/dl within 2 weeks of surgery
* Patients with contraindications to Angiotensin II including women who are pregnant or breastfeeding or have active coronary ischemia, mesenteric ischemia, limb ischemia, or high potassium (> 5.5 meq/L) while receiving Angiotensin II

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative acute kidney injury, atrial fibrillation | 28 days
  The primary endpoint will be measured by comparing the incidence of new-onset atrial fibrillation or acute kidney injury

SECONDARY OUTCOMES:
Hours on Vasopressors | 28 days
Total IVF | 28 days
ICU LOS | 28 days
Postoperative LOS | 28 days
Any major STS complication | 28 days
30-day mortality | 30 days
Cost | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland St. Joseph Medical Center, Towson, Maryland, United States

IPD SHARING:
Plan to Share IPD: No